CLINICAL TRIAL: NCT01242293
Title: Intrapartum Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0062-10-EMC; IH-1 (Other: 0062-10-EMC)
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Labor Stage, First; Labor Stage, Second
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.9% Saline with glucose 5% (Active Comparator): rate of infusion is 125cc/h
  Interventions: Other: 0.9% Saline with glucose 5%
- Ringer lactate (Active Comparator): rate of infusion is 250cc/h
  Interventions: Other: Ringer lactate
- Ringer lactate - Controls (Active Comparator): rate of infusion is 125cc/h
  Interventions: Other: Ringer lactate - Controls

INTERVENTIONS:
Other: 0.9% Saline with glucose 5% — intravenous hydration at a rate of 125 ml per hour during labor
  Arms: 0.9% Saline with glucose 5%
Other: Ringer lactate — intravenous hydration at a rate of 250 ml per hour during labor
  Arms: Ringer lactate
Other: Ringer lactate - Controls — intravenous hydration at a rate of 125 ml per hour during labor
  Arms: Ringer lactate - Controls

SUMMARY:
The purpose of this study is to determine that maternal hydration during labor with fluids containing glucose at a rate of 125 ml per hour does not affect the duration of labor compared to Ringer Lactate at a rate of 250 ml per hour.

DETAILED DESCRIPTION:
During labor it is a common practice that the parturient is fastening and having fluid replacement through intravenous hydration (IVH), the rational being to avoid aspiration of gastric content in a situation of need for urgent intervention and general anesthesia with tracheal intubation. It is acceptable to infuse 125 ml per hour of a physiological solution that does not contain sugar, but the volume is not adjusted to the weight of mother, the level of effort or relaxation she is experiencing and it may well be below the required amount. From studies in the field of sport medicine it is clear that the amount of fluid reaching the muscle has an impact on the efficiency of the muscle at the level of tissue and the level of personal achievement in sports. Only few studies dealt with the amount and contents of IVH during labor that will be sufficient and meet all physiologic requirements of the parturient and her fetus.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Gestational age 37-41 weeks
* Cervical dilatation 1-3 cm
* Vertex presentation
* Singleton

Exclusion Criteria:

* Diabetes
* Preeclampsia
* Intra uterine fetal growth restriction
* Duration of labor less than an hour
* Maternal chronic disease
* Maternal fever upon admission.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Length of time from enrollment until delivery | within the first 48 hours after delivery

SECONDARY OUTCOMES:
Mode of delivery | within the first 48 hours after delivery
Neonatal outcome | within the first 48 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Principal Investigator — Dep. OB/GYN, HaEmek Medical Center, Afula, Israel
Locations (1):
- Dep OB/GYN, HaEmek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Garmi G, Zuarez-Easton S, Zafran N, Ohel I, Berkovich I, Salim R. The effect of type and volume of fluid hydration on labor duration of nulliparous women: a randomized controlled trial. Arch Gynecol Obstet. 2017 Jun;295(6):1407-1412. doi: 10.1007/s00404-017-4381-1. Epub 2017 May 3. PMID 28470550